CLINICAL TRIAL: NCT02785198
Title: Passive Training as a Treatment for Diabetic Foot Ulcers: A Randomized, Single-blinded Clinical Trial of Wound Healing
Brief Title: Passive Training as a Treatment for Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to finalizing af phd project and fundings
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Tue Smith Jørgensen, Medical Doctor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-15008102
Record Dates: First submitted 2016-05-13; First posted 2016-05-27 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): A control group receiving standard wound treatment consisting of debridement, dressings, compression, offloading footwear and if necessary antibiotics.
- Passive training group (Experimental): An Intervention group doing passive exercise for 8 weeks in knee extensor machine, and receiving standard wound treatment consisting of debridement, dressings, compression, offloading footwear and if necessary antibiotics.
  Interventions: Device: Passive knee extensor machine

INTERVENTIONS:
Device: Passive knee extensor machine — The passive training machine, moves both legs from flexion to extension and back, 60 times per minute in 1 hour, 3 times per week. ROM is 60 degrees
  Arms: Passive training group

SUMMARY:
Overall project design: This PhD project involves a randomized study on diabetic individuals with healing resistant wounds, comparing the effect of passive movement of the lower limb with standard treatment of diabetic wounds.

How to effectively improve the condition of peripheral arterial disease is limited. The primary purpose of this study is to uncover whether passive movement of the lower limb will influence muscle oxygen demand and thereby increasing blood flow. An increase in muscle oxygen demand is likely to increase both blood flow rate and the number of capillaries, which would induce the healing of wounds, that were not previously possible.

The secondary purpose is to increase understanding of the pathophysiological processes in wound healing through the study of biochemical markers of vascularization, inflammation and stem cell recruitment in blood samples. Further on analyzing the skin and muscle biopsies of the number and quality of endothelial cells and Capillary density and to develop new quantifiable methods to evaluate wound healing in.

The project is a randomized trial, consisting of simple passive training to improve blood vessel function, increase the growth of the smallest blood vessels, thereby preventing ulceration and ultimately amputation.

DETAILED DESCRIPTION:
Background information

Diabetic foot ulcers are one of the most frequent and serious complication in diabetes mellitus. Despite attempts of prophylaxis*, only two-thirds of the diabetic foot ulcers eventually heal, and up to 15-20% will ultimately require a minor or major amputation (Major lower extremity amputation is defined as through or above the ankle joint, and minor amputations is below the ankle joint. The incidence of diabetes is growing, but the multifactorial causes of impaired healing of chronic diabetic ulcers are still not well understood.

The diabetic foot ulcers are known to reduce the quality of life for patients both psychically and psychologically and therefore further investigation in new treatment options is plausible. Current knowledge regarding how to improve the condition in the beginning phase of peripheral artery disease (PAD) is limited. Investigators know that high oxygen tension and perfusion of the limb as well as an adequate density of microvessels in the tissue, is essential to wound healing. Therefore, interventions that increase blood flow and promote microcirculatory growth are likely to be beneficial in the treatment of wound healing.

*Dressings, debridement, compression, clinical observation, antibiotics and glycemic control

It has been reported that passive training consisting of knee flexion/extension in a kinetic machine has a beneficial effect on up regulation of growth factors, remicrovascularization and improved blood flow. Høier et al described that passive movement of the leg induced a two-fold elevation in blood flow, elevation of angiogenic factors and initiates capillarization in skeletal muscle. All three factors are often impaired in the diabetic leg, which results in poor wound healing.

Due to the typical localization of the diabetic foot ulcers, this patient group is unable to exercise properly. Therefore will the investigators use a recent innovative model for the improvement of the limb microcirculation, developed at the Department of Nutrition, Exercise and Sports, University of Copenhagen, involving passive movement of the lower leg, for inducing increased blood flow and microcirculatory growth.

Rationale for the trial Diabetic patients have impaired wound healing due to multifactorial causes. The investigators know that high oxygen tension, and perfusion is essential to wound healing, and according to Høier et al's study, passive training can increase the perfusion and elevate proangiogenic factors in both young healthy males and peripheral artery disease (PAD) patients.

Null hypothesis:

1. Passive training does not lead to enhanced healing of diabetic foot ulcers.
2. Passive training of the lower limb does not affect perfusion of the trained limb.

Perspective:

This projects aim is to discover that passive training of the lower limb will increase the healing in diabetic foot ulcers. In addition, present a new treatment offer to diabetic patients with ulcers, who are not able to heal properly or perform active exercises. The investigators hope to see that the benefits of training and accelerated healing affect the PROM's.

Further on to present new knowledge of the specific molecular and functional changes that occur in the tissue during wound healing. This knowledge will be very important to improve our understanding of why ulcerations occur and why the tissue begins to decompose.

This is a prospective, randomized, single-blinded, parallel controlled design trial in subjects with diabetes mellitus investigating passive training as a treatment for the diabetic ulcer. The participants are randomized to either a control group or intervention.

The control group receiving standard wound treatment, and an intervention group receiving standard wound treatment, and passive training exercises for 8 weeks. The participants will be followed for 16 weeks or until clinical wound healing. All participants will receive standard wound care consisting of debridement, dressings, compression, offloading footwear and if necessary antibiotics The comparison groups should be as similar as possible as regard to important participant characteristics that might influence the response to the intervention. Therefore, a block randomization to ensure that equal numbers of participants with a characteristic thought to affect prognosis or response to the intervention, will be allocated to each comparison group.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
2. Diabetes mellitus according to the World Health Organisation (WHO) criteria (see http://www.who.int/diabetes/publications/en/ ) and a stable treatment treated in a period of 14 days prior to screening with insulin or an oral antidiabetic agent. Stable is defined as stable HBA1c.

4. Foot ulcer: size: diameter > 1cm. Duration of wound > 6 weeks Location: Full thickness skin defect distal to the malleoli.

5. Male or female, age >18 years at the time of signing informed consent. 6. Non-dementia diagnosis.

Exclusion Criteria:

1. Major infection; acute cellulitis, osteomyelitis or gangrene anywhere in the affected extremity.
2. Malignant disease
3. Major traumatic tissue damage.
4. Major lower extremity amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Wound healing change quantified by digital photo planimetry | Photos are taken at week 0 and 8
  The digital photo planimetry measurements are compared to the baseline measurement at week 0
The change in Wagner's wound classification. | week 0 and 8
  measurements at baseline are compared to week 8
The change in Wagner's wound classification. | week 3, 5 and 16
  The measurements at week 3, 5 and 16 are compared to the baseline week 0 and 8
Wound healing change quantified by digital photo planimetry | week 3, 5 and 16
  The measurements at week 3, 5 and 16 are compared to the baseline week 0 and 8

SECONDARY OUTCOMES:
Perfusion of the lower extremity. | week 0, 3, 5, 8 and 16.
  Quantified by measuring the blood flow in arteria femoralis (doppler)
Distal blood pressure measurement. | week 0 and 8.
  Includes skin perfusion test
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Hemoglobin mmol/L
Histological changes of the muscle tissue. | Week 0,5 and 8
  Analysed from muscle biopsies
Histological changes of the tissue composition in the edge of the wound. | Week 0,5 and 8
  Analysed from wound edge biopsy
Angiogenetic factors analysed from muscle biopsy | Week 0,5 and 8
  • Total RNA isolated from the muscle biopsies, and the mRNA content of VEGF, eNOS, MMP-2, MMP-9, TIMP-1, TIMP-2, Tie-2, ANG-1, ANG-2 determined by PCR
Dexa Scanning of the lower limb. | Week 0 and 8
  To measure the tissue composition change
Dexa Scanning of the lower limb. | Week 0 and 8
  To measure the bone mineral density change
Patient related outcome measurements (PROM's) | Week 0, 8 and 16
  Medical Outcome Study Short Form 36 (MOS SF36)
the change in 30 second chair stand test | Week 0 and 8
the change in maximum leg extension test | Week 0 and 8
Adverse events | Week 0, 3, 5, 8 and 16
Autonomic neuropathy | Week 0 and 8
  vagus device measurements at baseline and after 8 weeks
Distal blood pressure change measurement. | week 0 and 8
  Arm, ankle and toe pressure. The ankle brachial index (ABI) is calculated from measuring the arm and ankle systolic blood pressure.
Autonomic neuropathy | Week 0 and 8
  sudoscan measurements at baseline and after 8 weeks
Patient related outcome measurements (PROM's) | Week 0, 8 and 16
  the Euroqol five Dimensions questionnaire (EQ-5D)
Histological changes of the endothelial cells | 0,5 and 8
  analysed from muscle biopsies
Histological changes of the capillary density | 0,5 and 8
  Analysed from muscle biopsies
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Glycated HbA1c in mmol/mol
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Glucose in mmol/l
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  C-reactive protein in mg/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  leucocytes and differential count, in 10^9/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Thrombocytes in 10^9/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Sodium,mmol/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  potassium in mmol/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  eGlomerular filtration rate, mL/min/1,73 m^2
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Albumin g/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Creatinine, μmol/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Alanine Transaminase, U/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  Basic Phosphatase, U/L
The biochemical changes during wound healing, is assessed by biochemical markers in peripheral venous blood samples. | Week 0, 5 and 8
  YKL 40, μg/L

CONTACTS AND LOCATIONS:
Overall Officials: Tue Smith Joergensen, MD, Principal Investigator — Herlev and Gentofte Hospital, The Department of Orthopedics
Locations (1):
- Herlev Hospital, Herlev, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moxey PW, Gogalniceanu P, Hinchliffe RJ, Loftus IM, Jones KJ, Thompson MM, Holt PJ. Lower extremity amputations--a review of global variability in incidence. Diabet Med. 2011 Oct;28(10):1144-53. doi: 10.1111/j.1464-5491.2011.03279.x. PMID 21388445
- [Background] Tennvall GR, Apelqvist J, Eneroth M. Costs of deep foot infections in patients with diabetes mellitus. Pharmacoeconomics. 2000 Sep;18(3):225-38. doi: 10.2165/00019053-200018030-00003. PMID 11147390
- [Background] Baltzis D, Eleftheriadou I, Veves A. Pathogenesis and treatment of impaired wound healing in diabetes mellitus: new insights. Adv Ther. 2014 Aug;31(8):817-36. doi: 10.1007/s12325-014-0140-x. Epub 2014 Jul 29. PMID 25069580
- [Background] Hinchliffe RJ, Valk GD, Apelqvist J, Armstrong DG, Bakker K, Game FL, Hartemann-Heurtier A, Londahl M, Price PE, van Houtum WH, Jeffcoate WJ. A systematic review of the effectiveness of interventions to enhance the healing of chronic ulcers of the foot in diabetes. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S119-44. doi: 10.1002/dmrr.825. PMID 18442185
- [Background] Gary Sibbald R, Woo KY. The biology of chronic foot ulcers in persons with diabetes. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S25-30. doi: 10.1002/dmrr.847. PMID 18442179
- [Background] Jorgensen ME, Almdal TP, Faerch K. Reduced incidence of lower-extremity amputations in a Danish diabetes population from 2000 to 2011. Diabet Med. 2014 Apr;31(4):443-7. doi: 10.1111/dme.12320. Epub 2013 Oct 21. PMID 24111834
- [Background] Vogel TR, Petroski GF, Kruse RL. Impact of amputation level and comorbidities on functional status of nursing home residents after lower extremity amputation. J Vasc Surg. 2014 May;59(5):1323-30.e1. doi: 10.1016/j.jvs.2013.11.076. Epub 2014 Jan 7. PMID 24406089
- [Background] McDonald S, Sharpe L, Blaszczynski A. The psychosocial impact associated with diabetes-related amputation. Diabet Med. 2014 Nov;31(11):1424-30. doi: 10.1111/dme.12474. Epub 2014 May 24. PMID 24766143
- [Background] Jeffcoate WJ, Harding KG. Diabetic foot ulcers. Lancet. 2003 May 3;361(9368):1545-51. doi: 10.1016/S0140-6736(03)13169-8. PMID 12737879
- [Background] Pence BD, Woods JA. Exercise, Obesity, and Cutaneous Wound Healing: Evidence from Rodent and Human Studies. Adv Wound Care (New Rochelle). 2014 Jan 1;3(1):71-79. doi: 10.1089/wound.2012.0377. PMID 24761347
- [Background] Rasmussen BSB, Yderstraede KB, Carstensen B, Skov O, Beck-Nielsen H. Substantial reduction in the number of amputations among patients with diabetes: a cohort study over 16 years. Diabetologia. 2016 Jan;59(1):121-129. doi: 10.1007/s00125-015-3781-7. Epub 2015 Nov 22. PMID 26590707
- [Background] Hellsten Y, Rufener N, Nielsen JJ, Hoier B, Krustrup P, Bangsbo J. Passive leg movement enhances interstitial VEGF protein, endothelial cell proliferation, and eNOS mRNA content in human skeletal muscle. Am J Physiol Regul Integr Comp Physiol. 2008 Mar;294(3):R975-82. doi: 10.1152/ajpregu.00677.2007. Epub 2007 Dec 19. PMID 18094062
- [Background] Hoier B, Rufener N, Bojsen-Moller J, Bangsbo J, Hellsten Y. The effect of passive movement training on angiogenic factors and capillary growth in human skeletal muscle. J Physiol. 2010 Oct 1;588(Pt 19):3833-45. doi: 10.1113/jphysiol.2010.190439. PMID 20693292